CLINICAL TRIAL: NCT02723305
Title: Cardiometabolic Profiles of Pubertal Boys With Klinefelter Syndrome With or Without One Year of Exogenous Testosterone Treatment
Brief Title: Cardiometabolic Profiles of Boys With Klinefelter Syndrome
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 16-0248; UL1TR001082 (NIH)
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Klinefelter Syndrome; 47,XXY; Sex Chromosome Aneuploidy; XXY Syndrome
Keywords: Klinefelter syndrome; XXY; Sex chromosome aneuploidy; sex chromosome variation; hypogonadism; cardiometabolic; body composition; exercise capacity
MeSH Terms: conditions — Klinefelter Syndrome; Hypogonadism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Testosterone Naive: Boys with Klinefelter syndrome age 12-17 who are Tanner 3, 4, or 5. No exogenous testosterone exposure in the past 5 years
  Interventions: Other: No intervention
- Testosterone exposed: Boys with Klinefelter syndrome age 12-17 who are Tanner 3, 4, or 5.
  +topical testosterone treatment for >1 year
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
This study plans to learn more about how to measure the way the the body's energy system works in boys with Klinefelter syndrome, including the heart, lungs, muscles, and liver. This is important to know so that investigators understand how hormones and an extra X chromosome relate to diseases such as diabetes, extra weight gain, heart disease and liver diseases.

DETAILED DESCRIPTION:
Klinefelter syndrome (KS) is the most common chromosomal abnormality in males and is associated with primary gonadal failure in adolescence and a high morbidity and mortality from cardiovascular-related diseases (CVD) in adulthood. Recent studies in children and adolescent boys with KS have found a high prevalence of CVD risk markers, however the underlying mechanisms have not been explored. Our central hypothesis is that pubertal boys with KS have relative testosterone deficiency resulting in abnormal energy metabolism that predisposes them to later CVD, and that exogenous testosterone will modify these abnormalities.

In this study, investigators will measure markers of cardiometabolic risk in pubertal boys with KS.

ELIGIBILITY:
Inclusion Criteria:

* Male, 47,XXY karyotype (non-mosaic)
* Age 12-17 years
* Tanner stage 3-5 pubic hair
* T naïve group only: No exogenous androgen exposure within the past 5 years
* T exposed group only: currently on topical testosterone, with duration of treatment between 1-2 years.

Exclusion Criteria:

* Cognitive, psychiatric, or physical impairment resulting in inability to tolerate the study procedures
* MRI incompatible metal
* Diagnosis of type 1 or type 2 diabetes
* Hypertension greater than 140/90 mm/Hg at rest (would make exercise studies unsafe)
* Weight > 300 lbs (limit for DEXA)
* Testosterone treatment for <1 year or >2 years

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will enroll 10 youth with 47,XXY who will be subdivided into 2 groups:
  1. Testosterone naïve (no exogenous testosterone within the past 5 years)
  2. Testosterone exposed (topical testosterone treatment for at least 1 year but no more than 2 years) Most subjects will be recruited at the completion of a monitored, double-blind randomized controlled trial ongoing at our institution. Additional subjects may be recruited to meet enrollment goals.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
VO2 peak | baseline
  The primary outcome will be peak oxygen consumption (VO2 peak) during exercise on a bicycle ergometer

SECONDARY OUTCOMES:
Body composition | baseline
  Percent body fat by dual-energy x-ray absorptiometry
Liver fat | baseline
  Intrahepatic fat by abdominal magnetic resonance imaging
Muscle mitochondrial metabolism | baseline
  Rate of mitochondrial phosphorylation by 31-phosphorus magnetic resonance spectroscopy of the calf muscles
Insulin sensitivity | baseline
  oral disposition index with Glucola

CONTACTS AND LOCATIONS:
Overall Officials: Shanlee M Davis, MD, Principal Investigator — University of Colorado/Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis SM, DeKlotz S, Nadeau KJ, Kelsey MM, Zeitler PS, Tartaglia NR. High prevalence of cardiometabolic risk features in adolescents with 47,XXY/Klinefelter syndrome. Am J Med Genet C Semin Med Genet. 2020 Jun;184(2):327-333. doi: 10.1002/ajmg.c.31784. Epub 2020 Jun 16. PMID 32542985